CLINICAL TRIAL: NCT02692872
Title: Screening for Alpha Globin Deletions
Brief Title: Screening for Alpha Thalassemia in Healthy Volunteers
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160065; 16-I-0065
Record Dates: First submitted 2016-02-25; First posted 2016-02-26 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-06-16

CONDITIONS: Alpha Thalassemia
Keywords: Alpha Thalassemia; Double Deletion
MeSH Terms: conditions — alpha-Thalassemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: We plan to perform genetic screening of up to 2,000 individuals of African ancestry, an ethnic group with a high prevalence of alpha thalassemia.

SUMMARY:
Background:

Alpha thalassemia is a blood disorder. It is caused by genetic deletions. Part of the DNA is missing from a group of genes called alpha globin. Alpha thalassemias are some of the most common genetic deletions. We are testing for alpha thalassemia trait. Alpha thalassemia trait is when someone has only two out of the normal four alpha globin genes. In some people, they lead to no symptoms. Others have changes that lead to disease, including mild anemia. Researchers want to learn more about alpha thalassemia and blood vessels. This may allow them to develop new treatments for blood diseases such as sickle cell disease.

Objective:

To better understand how alpha globin deletions in healthy people affect blood vessels.

Eligibility:

Healthy volunteers ages 18-39 who self-report African ancestry.

Design:

Participants will provide a one-time saliva sample. This can be by mail, in-person at a study event, or at NIH.

Participants will get a small kit to collect their saliva sample. The kit has easy instructions. The sample does not need to be put in the refrigerator.

Participants will spit a small amount of saliva (less than half a teaspoon) into a collection tube.

Participants will close the funnel lid tightly, and then unscrew the funnel lid from the tube. They will then close the tube tightly with the small cap provided and shake the tube for 5 seconds.

Participants will place the tube in the provided envelope and mail it to NIH. The specimen will be stored and processed in the lab.

Participants may be invited to participate in more research studies, whether or not researchers find that they have alpha thalassemia trait.

DETAILED DESCRIPTION:
Many of the complications of sickle cell disease, such as stroke, kidney damage, skin ulceration,pulmonary hypertension, and cardiac hypertrophy are prevented, delayed or reduced by inheritance of one of more deletions of the alpha globin genes. Our long-term research goal is to understand how deletions of alpha globin protect against the vascular complications of sickle cell disease.

Deletions of alpha globin are common and found in approximately 5% of the world s population.They are especially common among Africans and people of African ancestry, as well as in India, China, and the Pacific Islands, where prevalence can range from 5 - 80%. A single deletion has little effect on the red blood cell, but two deletions can give rise to alpha thalassemia, a mild microcytic anemia. Patients with sickle cell disease who have two alpha globin deletions tend to have a higher hemoglobin level, smaller red blood cells, and a lower fraction of circulating reticulocytes - consistent with decreased hemolysis and red cell turnover. They also have a lower number of dense or irreversibly sickled cells. These changes might explain why alpha globin deletions reduce the severity of sickle cell disease.

However, a novel function for alpha globin as a regulator of endothelial nitric oxide (NO) has recently been identified that raises new questions about how alpha globin deletions protect against sickle cell disease. We hypothesize that individuals with two alpha globin deletions will have decreased gene expression and protein levels of alpha globin in vascular endothelium, permitting more NO to diffuse across the myoendothelial junction, compared to individuals who have all four alpha globin genes intact. In this protocol we will screen healthy volunteers to identify those with two alpha globin deletions; these individuals as well as matched controls will be referred to a separate protocol to undergo studies of vascular endothelial function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject report of the following:

1. Age 18 - 39
2. Self-report of African ancestry
3. Willingness and legal ability to give and sign informed study consent

EXCLUSION CRITERIA:

There are no exclusion criteria for this screening protocol

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All subjects ages 18 through 39 will be considered for the protocol. We have excluded anyone age 40 and older in order to avoid confounders of older age and cardiovascular disease in asymptomatic subjects. No subject will be excluded from participation based on gender. Subjects will be enrolled based on self-report of African ancestry given the higher prevalence of the genetic mutation in these populations.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify Presence of Double Alpha Globin Deletions in Healthy Volunteers. | Ongoing
  As this is not a treatment protocol, there is no primary endpoint. The primary objective is to identify presence of double alpha globin deletions in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Amy P Ruhl, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The IPD is not required for non-interventional, non-clinical trials.

REFERENCES:
- [Background] Piel FB, Weatherall DJ. The alpha-thalassemias. N Engl J Med. 2014 Nov 13;371(20):1908-16. doi: 10.1056/NEJMra1404415. PMID 25390741
- [Background] Embury SH, Dozy AM, Miller J, Davis JR Jr, Kleman KM, Preisler H, Vichinsky E, Lande WN, Lubin BH, Kan YW, Mentzer WC. Concurrent sickle-cell anemia and alpha-thalassemia: effect on severity of anemia. N Engl J Med. 1982 Feb 4;306(5):270-4. doi: 10.1056/NEJM198202043060504. PMID 6172710
- [Background] Straub AC, Lohman AW, Billaud M, Johnstone SR, Dwyer ST, Lee MY, Bortz PS, Best AK, Columbus L, Gaston B, Isakson BE. Endothelial cell expression of haemoglobin alpha regulates nitric oxide signalling. Nature. 2012 Nov 15;491(7424):473-7. doi: 10.1038/nature11626. Epub 2012 Oct 31. PMID 23123858
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0065.html